CLINICAL TRIAL: NCT03034980
Title: Influence of Training Intensity on Exercise Capacity and Risk Profile in Coronary Artery Disease
Brief Title: Influence of Training Intensity in Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, prof. dr., Hasselt University
Other Study IDs: PD-VG-01
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Workload

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD) patients: Patients with proven coronary artery disease, who underwent the full cardiac revalidation program at Jessa Hospital from 10-1-2013 till 12-9-2016.
  Interventions: Other: Training intensity (workload) during ergospirometry

INTERVENTIONS:
Other: Training intensity (workload) during ergospirometry — The reached workload (W) during each training is noted during 12 weeks of rehabilitation. The relative intensity is expressed as a percentage of VT1 and VT2.

SUMMARY:
Coronary artery disease (CAD) is associated with high mortality worldwide. Narrowing of the coronary arteries can cause an acute myocardial infarction. Patient with cardiac ischemia are often treated with percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG). Following hospitalisation, the patients are offered to attend a classical rehabilitation program with moderate exercise intensity. Current exercise program for cardiac rehabilitation has proven to reduce cardiovascular risk factors 1. Is it possible to improve the exercise capacity and risk profile even more if the exercise program includes more vigorous training? The program starts one week after the cardiac incident (AMI, PCI or CABG) and takes 12 weeks to complete. Patients with heart failure and valvular disease are excluded. First ventilatory threshold (VT1) and second ventilatory threshold (VT2) are determined during cycloerometry. VT2 reflects aerobic-anaerobic transition and therefore the aerobic functional capacity2. Exercise load reached at VT2 is used to determine the training load during rehabilitation.

The research goal is to investigate the influence of training intensity on the exercise capacity and risk profile of CAD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myocardial infarction (AMI), who underwent a percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG). The 12-week program must be completed.

Exclusion Criteria:

* Patients with heart failure (HFpEF and HFrEF with ejection fraction ≤40%) and valvular heart disease.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proven coronary artery disease, who underwent the full cardiac revalidation program at Jessa Hospital from 10-1-2013 till 12-9-2016.
Sampling Method: Probability Sample
Enrollment: 343 (Estimated)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
exercise capacity | up to week 12
  The primary endpoint is the relationship between the actual training load (W) and exercise capacity (VO2max) obtained at the end of the rehabilitation.

SECONDARY OUTCOMES:
cardiovascular risk profile | up to week 12
  The secondary endpoint is the relationship between relative training load and the cardiovascular risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Kaatje Goetschalckx, MD, Principal Investigator — Catholic University Leuven, Belgium
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No